CLINICAL TRIAL: NCT04115969
Title: Outcome After Non-invasive Ventilation - an Observational Study at the Intensive Care Unit at Sundsvall Hospital.
Brief Title: Outcome After Non-invasive Ventilation.
Status: Completed | Type: Observational
Sponsor: Jakob Wallden (Other Government)
Responsible Party: Sponsor-Investigator, Jakob Wallden, Senior Lecturer, Consultant Anesthesiologist, MD, PhD., Västernorrland County Council, Sweden
Organization: Västernorrland County Council, Sweden (Other Government)
Other Study IDs: NIV-SUNDSVALL
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Insufficiency
Keywords: non-invasive ventilation; critical care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with non-invasive ventilation

SUMMARY:
The study is an exploratory retrospective observational study with the aim to describe outcome fo the cohort of patients that receive non-invasive ventilation at an intensive care unit.

Main research questions are:

* Characteristics of the cohort.
* The course for the patients at the ICU.
* ICU-mortality and 30-day mortality
* Amount of patients with limitations of care.
* Factors associated with mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Non invasive ventilation
* Admitted to Sundsvalls ICU during 2018

Exclusion Criteria:

* Below 18 years age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Sundsvalls intensive care unit treated with non-invasive ventilation.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Patient characteristics | At the day of admission to the ICU - 1 day
  Age, gender, comorbidities, indications for respiratory support, BMI, limitations of care.
ICU-mortality | Patients will be followed during their ICU-stay - estimated to be 1 to 60 days.
  Death occuring during ICU stay
30-day mortality | 30 days from admission to ICU
  Death within 30 days after ICU admission

SECONDARY OUTCOMES:
Factors associated with mortality | 30 days from admission to ICU
  Evaluate patient and ICU-factors and relation to mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Svensk, MD, Principal Investigator — Västernorrland county council (Region Västernorrland)
Locations (1):
- Västernorrland County Council / Sundsvall Hospital, Sundsvall, X, Sweden